CLINICAL TRIAL: NCT03577067
Title: Complicated Outcome Prediction After Liver Resection: the Role of Renal Resistive Index
Brief Title: Complicated Outcome Prediction After Liver Resection
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, MD, PhD, FACS, Humanitas Clinical and Research Center
Other Study IDs: CE Humanitas 100/15
Record Dates: First submitted 2018-05-28; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients submitted to liver resection: Patients underwent liver resection for primary and secondary disease
  Interventions: Procedure: Liver resection for primary and secondary disease

INTERVENTIONS:
Procedure: Liver resection for primary and secondary disease — Liver resection in parenchyma-sparing setting for primary and secondary disease

SUMMARY:
Although mortality after liver surgery reduced during the last three decades to less than 2%, post-operative course is still complicated in a range of 20-50% of cases.The identification of one or few factors which could detect the real risk of complicated post-operative outcome, may help anesthesiologist to decide whether admit a patient to ICU or not.The primary aim of this study was to evaluate whether RRI, alone or along with other items, can predict post-operative complication after hepatic resection.

ELIGIBILITY:
Inclusion Criteria:

Patients resectable and affected by primary and secondary liver disease

Exclusion Criteria:

Subjects affected by kidney disease and/or cirrhosis and pregnant patients were excluded from the trial. Patients who should have needed nephrectomy during the operation would be also excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients resectable and affected by primary and secondary liver disease
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
renal resistive index (RRI) | up to 7 days after surgery
  the association between RRI and occurrence of hepatic complications during the first postoperative week.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Torzilli, MD, PhD, Principal Investigator — Humanitas University

IPD SHARING:
Plan to Share IPD: No